CLINICAL TRIAL: NCT04749524
Title: Otoacoustic Emission Suppression in Clinical Populations
Brief Title: Otoacoustic Emission Suppression Study
Status: Completed | Type: Observational
Sponsor: Intelligent Hearing Systems (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: MOCR
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Newborns: Newborns from NICU or well-baby nursery.
  Interventions: Diagnostic Test: Medial-Olivocochlear Reflex (MOCR) Strength Measurement
- Newborn Hearing Screening Results: Newborns identified as having difficulty passing newborn hearing screening.
  Interventions: Diagnostic Test: Medial-Olivocochlear Reflex (MOCR) Strength Measurement
- Adults with Normal Hearing: Adults with normal hearing thresholds.
  Interventions: Diagnostic Test: Medial-Olivocochlear Reflex (MOCR) Strength Measurement
- Participants with Neural Hearing Loss: Participants, children and adults, with neural hearing loss.
  Interventions: Diagnostic Test: Medial-Olivocochlear Reflex (MOCR) Strength Measurement

INTERVENTIONS:
Diagnostic Test: Medial-Olivocochlear Reflex (MOCR) Strength Measurement — Otoacoustic emissions (OAE) will be recorded using an ear probe with and without an efferent Medial-Olivocochlear Reflex (MOCR) elicitor.

SUMMARY:
The focus of this project is on a physiologic auditory response called the Medial Olivocochlear Reflex (MOCR) that assesses peripheral neural function. While neural hearing loss is a significant auditory disorder in patients of all ages, more than 50% of newborn infants are screened with a technology that is not sensitive to abnormalities in neural function. The development of a time-efficient and sensitive test system to assess the MOCR will provide significant benefit to infants and patients of all ages with neural deficits who would otherwise go undetected.

DETAILED DESCRIPTION:
The objective of this study is to develop an optimized hearing testing method using otoacoustic emissions, that can be used to efficiently assess peripheral neural function (including retrocochlear disorders) using the medial olivocochlear reflex (MOCR). Measuring neural function via the MOCR. This reflex has been shown to be abnormal in patients with neural disorders. The focus of this project will be the development of a screening method that incorporates OAE screening and measurement of the MOCR in the same test procedure. The target population in the proposed research is infants, particularly those in environments where auditory brainstem response (ABR) screening is not performed routinely. Addition of the MOCR to screening where ABR is not performed will address the shortcoming of OAE screening which misses neural forms of hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Normal middle-ear function
* Present TEOAEs.

Exclusion Criteria:

* Atresia or other external ear abnormalities not allowing recording of OAEs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and newborns with normal middle ear function and no external ear abnormalities such as atresia
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Hood, PHD, Study Director — Vanderbilt University Medical School; Rafael E Delgado, PHD, Principal Investigator — Intelligent Hearing Systems Corp
Locations (1):
- Vanderbilt University Medical School, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
The results from the project will be shared by presenting results at scientific conferences and publishing results in scientific journals. In addition, a de-identified database containing subject gender, age at recording, raw MOCR recordings, recording parameters and spectral analysis parameters will be maintained. The data will be shared with other centers conducting similar research under appropriate IRB approval.

REFERENCES:
- [Background] Hood LJ, Berlin CI, Bordelon J, Rose K. Patients with auditory neuropathy/dys-synchrony lack efferent suppression of transient evoked otoacoustic emissions. J Am Acad Audiol. 2003 Aug;14(6):302-13. PMID 14552424
- [Background] Hood LJ, Berlin CI, Hurley A, Cecola RP, Bell B. Contralateral suppression of transient-evoked otoacoustic emissions in humans: intensity effects. Hear Res. 1996 Nov 1;101(1-2):113-8. doi: 10.1016/s0378-5955(96)00138-4. PMID 8951438
- [Background] Abdala C, Mishra S, Garinis A. Maturation of the human medial efferent reflex revisited. J Acoust Soc Am. 2013 Feb;133(2):938-50. doi: 10.1121/1.4773265. PMID 23363111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the general Vanderbilt University community and surrounding area population (children 6 years and older and adults with normal hearing), audiology clinics (infant, children 6 years and older, and adults with hearing loss), and infants at the Newborn (Well-Baby) Nursery and the Neonatal Intensive Care Unit (NICU) at the Vanderbilt Monroe Carell Jr. Children's Hospital (VCH).
Groups:
- Newborns: Newborns
- Newborn Hearing Screening: Newborns identified as having difficulty passing newborn hearing screening.
- Participants With Neural Hearing Loss: Participants having a neural hearing loss.
Period: Overall Study
Arm/Group | Newborns | Newborn Hearing Screening | Adults With Normal Hearing | Participants With Neural Hearing Loss
Started | 166 | 22 | 45 | 3
Completed | 166 | 22 | 45 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With Neural Hearing Loss: Participants with neural hearing loss.
- Total: Total of all reporting groups
Arm/Group | Newborns | Newborn Hearing Screening Results | Adults With Normal Hearing | Participants With Neural Hearing Loss | Total
Number analyzed (Participants) | 166 | 22 | 45 | 3 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.014 (0.049) | 0.072 (0.047) | 29.23 (6.34) | 15.67 (6.43) | 4.77 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 6 | 42 | 1 | 128
  Male | 87 | 16 | 3 | 2 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 3 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 26 | 0 | 3 | 0 | 29
  White | 115 | 18 | 39 | 3 | 175
  More than one race | 7 | 1 | 0 | 0 | 8
  Unknown or Not Reported | 14 | 3 | 0 | 0 | 17
Region of Enrollment [Number; unit: participants]
  United States | 166 | 22 | 45 | 3 | 236

OUTCOME MEASURES:

1. Primary Outcome: Otoacoustic Suppression Measure
Description: The decibel (dB) Sound Pressure Level (SPL) of the otoacoustic emission (OAE) response will be measured when recorded with and without an elicitor. The dB difference between the two measures, the OAE suppression, is used to calculate the Medial-Olivocochlear Reflex (MOCR) Strength. The elicitor is presented using a temporally separated and spectrally separated method, resulting in the two MOCR Strength measurements reported.
Time Frame: Within 48 hours of measurement
Population: Results from subjects with high ambient or physiological acoustic noise were excluded. For the Newborn Hearing Screening group, only the spectrally separated MOCR Strength method was used due to time limitations.
Measure: Mean (Standard Deviation); unit: dB - Unitless Difference in dB SPL
Arm/Group | Newborns | Newborn Hearing Screening Results | Adults With Normal Hearing | Participants With Neural Hearing Loss
Number analyzed (Participants) | 45 | 22 | 23 | 3
dB - Unitless Difference in dB SPL
  MOCR Strength (Spectrally Separated Method) | 1.95 (1.41) | 1.33 (1.22) | 2.48 (1.74) | 0.36 (0.32)
  MOCR Strength (Temporally Separated Method): number analyzed (Participants) | 11 | 0 | 23 | 3
  MOCR Strength (Temporally Separated Method) | 1.57 (2.22) |  | 1.79 (1.10) | 0.35 (0.18)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Newborns | Newborn Hearing Screening Results | Adults With Normal Hearing | Participants With Neural Hearing Loss
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/22 | 0/45 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/22 | 0/45 | 0/3
Other Adverse Events (participants affected / at risk) | 0/166 | 0/22 | 0/45 | 0/3

LIMITATIONS AND CAVEATS:
The measurement of the medial-olivocochlear reflex (MOCR) using otoacoustic emissions (OAEs) as the assay requires that participants have present OAEs. Thus, participants who do not have OAEs, which can be due to middle-ear problems or sensorineural hearing loss affecting cochlear active processes, would not be candidates for this type of measure. OAEs are low amplitude signals that are generated from the inner ear. Therefore, a quiet participant and quiet test environment are required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04749524/Prot_SAP_ICF_000.pdf